CLINICAL TRIAL: NCT04468451
Title: Does Dosage Matter: A Randomized Controlled Trial of ride-on Car Training With a Standing Posture to Enhance Social-mobility Function and Motivation in Toddlers With Motor Disabilities
Brief Title: Does Dosage Matter: Ride-on Cars to Enhance Social-mobility Function and Motivation in Toddlers With Motor Disabilities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Hsiang-Han Huang, Associate Professor, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201802038A3
Record Dates: First submitted 2020-07-08; First posted 2020-07-13 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Mobility Limitation
Keywords: toddlers with disabilities; modified ride-on cars; social-mobility; mastery motivation; physical activity; family participation
MeSH Terms: conditions — Mobility Limitation; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ROC-48 group (Experimental): The participant's performance is indicative of the extent to which early power mobility training is feasible for 1 to 3 years old and diagnosed as motor delay. Parents/caregivers and the occupational therapist will be responsible for ride-on car with a standing posture training. The dosage will be 48 hours for a total of 12-week intervention.
  Interventions: Behavioral: A 48-hour ROC training program with a standing posture
- ROC-24 group (Active Comparator): The participant's performance is indicative of the extent to which early power mobility training is feasible for 1 to 3 years old and diagnosed as motor delay. Parents/caregivers and the occupational therapist will be responsible for ride-on car with a standing posture training. The dosage will be 24 hours for a total of 12-week intervention.
  Interventions: Behavioral: A 24-hour ROC training program with a standing posture
- Control group (Active Comparator): The participant's performance is indicative of the extent to which early power mobility training is feasible for 1 to 3 years old and diagnosed as motor delay. The participant's clinical occupational therapist will be responsible for the regular therapy. The dosage will be their regular dosage for a total of 12-week intervention.
  Interventions: Behavioral: A regular therapy program without receiving any ROC training

INTERVENTIONS:
Behavioral: A 48-hour ROC training program with a standing posture — The 2-hour training session is composed of two 30-minute driving sessions and two 25-minute natural play sessions, with a 10-minute break. Every week's treatment program will be before planned and adjusted by the therapist and the caregivers through discussion and clinical observation of participant's performance in the previous session. Training will concentrate on building the concept of casual-effect on the switch and car motion, goal-oriented driving in a hospital, and upper limb use in functional tasks with driving and hand use in functional tasks for exploration in natural play session.
  Arms: ROC-48 group
Behavioral: A 24-hour ROC training program with a standing posture — The 1-hour training session is composed of a 30-to-35-minute car play and a 25-minute natural play. Every week's treatment program will be before planned and adjusted by the therapist and the caregivers through discussion and clinical observation of participant's performance in the previous session. Training will concentrate on building the concept of casual-effect on the switch and car motion, goal-oriented driving in a hospital, and upper limb use in functional tasks with driving and hand use in functional tasks for exploration in natural play session.
  Arms: ROC-24 group
Behavioral: A regular therapy program without receiving any ROC training — The regular therapy group will be an active control group without receiving any additional training. The training dosage will be their own therapy, including occupational, physical and speech therapy. They will continue their regular therapy, including physical, occupational and speech therapy. The general propose of the training is to improve the developmental scales, mobility, socialization and upper limb use in functional tasks.
  Arms: Control group

SUMMARY:
Modified ride-on toy cars (ROCs) have been viewed as one Maker Movement and become an innovative, alternative option to enhance independent mobility and socialization in young children with disabilities in the recent years. To increase the applicability of this novel intervention, this study proposes a modified ROC-training program with a less-intensive dose which may be an effective and a more feasible protocol for clinical therapists and caregivers to implement.

The three purposes of this study are: 1) to compare the effectiveness of different dosages of ROC training with a standing posture on social-mobility function, mastery motivation and physical activity in toddlers with motor disabilities; 2) to determine the optimal dosage of ROC training with a standing posture that is needed to enhance social-mobility function, mastery motivation and physical activity in toddlers with motor disabilities; and 3) to examine the effects of different dosages of ROC training with a standing posture on the ICF functioning levels, family perceptions and participation.

Based on the power analysis from the preliminary results of our RCT study, the investigator will recruit 45 children with disabilities who are between 1 to 3 years old and diagnosed as motor delay. They will be randomly assigned to one of the following three groups: a 48-hour ROC training program with a standing posture (ROC-48) (n=15), a 24-hour ROC training program with a standing posture (ROC-24) (n=15), and a regular therapy program without additional training (n=15). The whole study duration will be 24 weeks, including 12-week intervention and 12-week follow-up. The ROC-48 and ROC-24 programs will include 2 sessions/per week, each session for 1 hour (ROC-24) or 2 hours (ROC-48) training. All participants will continue their regular therapy during the whole study. Standardized assessments are provided for a total three times, including the time before and after the intervention and in the end of the follow-up phase. Assessments include social mobility, mastery motivation, behavioral coding, body function, family perception and participation. The use of modified toy cars with different dosages will provide the family and therapists a set of novel, alternative ways to increase family participation and facilitate development in toddlers with disabilities, depending on children's and family's needs.

DETAILED DESCRIPTION:
There is increasing evidence of early power mobility training in recent years, which focuses on the outcomes of motivation and socialization by using standardized measurements, including the Dimensions of Mastery Questionnaire (DMQ), the pediatric evaluation of disability inventory (PEDI) and its' computer adaptive test. These studies showed the use of PMDs might increase the child's independent mobility and motivation to master interpersonal tasks and result in positive changes on psychosocial functioning. Previous studies have determined the feasibility of using a modified ride-on car (ROC) as an alternative, novel option for early mobility training to improve independent mobility and socialization in children aged younger than 3 years. Of note is that this technology-focused do-it-yourself (DIY) movement has provided concrete solutions for children with disabilities, which emphasizes "learning by doing" and is called "the Maker Movement". Awori and Lee has viewed the process of modifying the ROCs and applying relevant training as one Maker Movement. Due to the participatory model of innovation, there are over 60 workshops worldwide that have built approximately 5000 ride-on toy cars. In addition to this universal trend of hands-on practice for health innovation, the use of ROCs may result in the significant improvements in motivation and physical activity in young children with motor disabilities.

Kenyon and colleagues reported that pediatric occupational therapists and physical therapists in Canada and the USA recognized the potential benefits of applying power mobility training in young children who have mobility impairments. In addition, almost all therapists agreed or strongly agreed that time and practice were equally as important as a child's abilities when applying power mobility training. However, 69% of these therapists never or seldom provided these types of experiences to children in their practice. The amount and type of practice may play an important role while making the clinical decision. Based on the increased evidence for children with motor disabilities in the past 10-15 years, researchers have suggested that the type of treatment may matter less than the amount of treatment (dosage). The idea of providing an intervention at an amount of greater than standard care has generally been conceptualized with the terms "intensity or intensive treatment". Up to now, several ROC studies have suggested intensive dose of therapy may be effective on improving social-mobility function and mastery motivation. Although the participants were able to complete the 12-week training, the caregivers felt it may be difficult to implement such program in their clinical settings. Our previous pilot results have shown that 85% of the caregivers preferred a 1-hr program than a 2-hr program due to the family resources and geographical concerns. The current ROC training program typically involves long length (9-12 weeks), high frequency (2 sessions per week) and duration (2 hours per session). However, the high frequency and duration may not be a feasible protocol for therapists and caregivers. In addition, there is no study comparing the same type of ROC training at contrasting doses and therefore could not address the relative effectiveness of different doses of therapy. A further study with the comparison of different doses of training may help to determine the optimal program for enhancing social-mobility and psychosocial functions in toddlers with motor disabilities.

It is important to consider the clients' needs and incorporate the suggestions into the training protocol based on the evidence. To integrate the caregivers' feedback and increase the applicability of the ROC training program, the investigator further propose a modified program of using the ROC with less-intensive doses, i.e., a 1 hour session of 30-to-35-minute standing-driving for exploration and 25-minute natural play for exploration and skills training. The investigator assume the less-intensive dose of the ROC training will also have positive effects on social-mobility function and other ICF levels due to the sufficient amount of practice suggested by previous evidence (at least 20 to 60 min. moderate to vigorous intensity/per session, 2 sessions/per week). A 3-group comparison design of different doses of ROC training with a standing posture may provide us a complete examination on the topic of dose-response effect on mobility and psychosocial function in toddlers with disabilities. In this study, the investigator will modify the ride-on toy car (standing style) for toddlers with disabilities for the use in the public spaces in the university for 12 weeks based on our previous RCT study. This RCT will compare the improvements of social-mobility function, mastery motivation and physical activity resulting of different dosages for the ROC use with a standing posture. A control group which receives no ROC training and only involves regular therapy will be applied as an active control group.

The specific aims of this study are: 1) to compare the effectiveness of different dosages of ROC training with a standing posture on social-mobility function, mastery motivation and physical activity in toddlers with motor disabilities; 2) to determine the optimal dosage of ROC training with a standing posture that is needed to enhance social-mobility function, mastery motivation and physical activity in toddlers with motor disabilities; and 3) to examine the effects of different dosages of ROC training with a standing posture on the ICF functioning levels, family perceptions and participation.

Study Design: A randomized, multiple group pretest-posttest control group design will be applied.62 Three groups will be involved in this novel project: the dosage of a 48-hour ROC training program with a standing posture (ROC-48), the dosage of a 24-hour ROC training program with a standing posture (ROC-24), and a regular therapy program without receiving any ROC training (control). The participants will be randomly assigned to one of the 3 groups by using a computer program (Research Randomizer Form www.randomizer.org). The study duration for each participant is 24 weeks, including 12-week intervention and 12-week follow-up.

Recruitment: The participants will be recruited from self-referrals, health care practitioners, or the hospitals in Taipei or Taoyuan where toddlers with motor delays are receiving outpatient rehabilitation. The research team will contact the parent/guardian to explain study details and provide them the opportunity to ask questions. Parents will receive a letter detailing the procedure; children of parents/guardians who provide informed consent will participate in the study.

Procedure: Before the pre-intervention assessments, the research team will modify the car's seat and acceleration to the hand switch-driven. After modifications, they will receive pre-intervention measurements, including developmental assessments, behavioral videotaping and self-developed questionnaires. These assessments will occur on three occasions: before and after the 12-week intervention (T1 & T2) and the end of the 12-week follow-up phase (T3). During the 12-week intervention, the social-mobility behaviors for the 2 ROC training groups will also be videotaped by the research team for 1 hour during one session/per week at the university. In addition, participants will wear three accelerometers on their wrists and right hip to monitor the minutes of exercise, postural change, activity counts and energy expenditure for exploration during one training session/each week for 12 weeks. An activity log used in the previous studies will also be applied to record the driving and play duration, driving locations, and the caregiver's feedback on the training program every week.

Intervention: The research team will ask caregivers to identify goals (before intervention), and measure progress using goal-attainment scaling (GAS) at T1 and T2 time points for the 2 ROC training groups. An independent licensed occupational therapist who will not involve the administration of assessments will provide the intervention with the caregivers. The training principles are similar to those applied in our previous studies of ROC training in various environments. To record the total driving time, locations, and caregivers' feedback regarding training, an activity log will be used for each week. All groups will continue their regular therapy from their own therapists throughout the 24-week duration of the study, including physical therapy, occupational therapy, and speech therapy. The research team do not provide regular therapy during the study.

On licensed, independent OT will provide the ROC training programs for the two ROC training groups. The ROC-48 will receive the program in the university for 2 hours/per session, 2 sessions/per week for a total of 12-week intervention. For the ROC-24 group, the participants will have a 30-to-35-minute car play and a 25-minute natural play and the frequency is 2 sessions/per week for a total of 12 weeks. The training programs for the two ROC training groups will be based on the ecological and dynamic systems theory. All the programs will be discussed by the family, the treating therapist and the research team. The program for the control group will only involve their regular therapy provided by their own clinical therapists.

Follow-up: This period will involve a 12-week phase following the above treatment programs; during this time no treatment programs will be delivered to the participants except for their own regular therapy.

Data Reduction and Analysis: Social-mobility measures will be obtained every week during the intervention phase, including the simultaneous co-occurrence of self-directed locomotion and direct adult interaction, and operationalized as number of minutes observed. All data records will exclude names to provide anonymity of the participant. Two independent coders will code all the videotapes related to social-mobility and mastery motivation performances. In addition, they will determine the physical activity for exploration by combining the data from activity monitors and the videotapes. All the coding criteria of social-mobility and mastery motivation are established based on the previous studies.

Descriptive statistics including frequency, means, standard deviations, as well as nonparametric data medians and interquartile ranges will be calculated. Kolmogorov-Smirnov will be used to examine whether the data follows a normal distribution. To compare the baseline characteristics of the 3 groups, one-way ANOVA (for data with normal distribution) and Kruskal-Wallis test (for data with non-normal distribution) will be conducted. If there is a significant difference among the 3 groups, the specific baseline characteristics will be analyzed and further determined as the co-variate for the subsequent analysis, e.g., regular therapy. Data will be analyzed based on an intention-to-treat analysis. A repeated measures analysis of variance (group [3] × time [3]) will be employed to evaluate the treatment effects on the primary and secondary outcomes among the 3 groups at T1, T2, and T3, followed by a post-hoc analysis using Bonferroni test to determine between which groups the differences occur. SPSS 20.0 (SPSS Inc. Chicago, Illinois, USA) will be used for statistical analysis. Significance level will be set at p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* 1. motor delays that resulted in motor impairments that prevented independent walking (standard deviation (SD) < -1.5, assessed by the Chinese Child Development Inventory (CCDI) via a pediatric physician) 2. can stand independently for two seconds or to tolerate standing with support for 10 minutes 3. can reach for objects/toys with either one or two hands 4. the height is between 69 to 103 cm and the weight is between 7-18 kg 5. parents are able to provide consent for their child's participation in training programs

Exclusion Criteria:

* 1. children with severe sensory impairments such as blindness, deafness 2. the height is not between 69 to 103 cm and the weight is not between 7 to 18 kg 3. parents/caregivers are not able to make a time commitment for the training phase

Ages: 12 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 13 (Actual)
Dates: Start 2020-08-05 (Actual); Primary Completion 2022-05-05 (Actual); Study Completion 2022-07-29 (Actual)

PRIMARY OUTCOMES:
Change from baseline in General Mobility and Social Development at 12 weeks and 24 weeks as assessed by the Cinese version of Pediatric Evaluation of Disability Inventory (PEDI) | Assessment will occur 3 times during the whole study, including the first and last week of the 12-week intervention, and the end of the 12-week follow-up phase
  EDI is a set of tests for children from 8 months to 6 years old. The PEDI quantified self-care, mobility, and social functions. The PEDI is especially useful for tracking changes in functional skills.
Social-Mobility Performance | The socialization behaviors will be followed for the duration of implementing the intervention phase, an expected average of 12 weeks
  Every week during the intervention phase, the first 1 hour session will be recorded. The social-mobility behavior is defined as the simultaneous co-occurrence of self-directed locomotion and direct adult interaction, and operationalized as number of minutes observed.

SECONDARY OUTCOMES:
Change from baseline in Body Function/Structure at 12 weeks and 24 weeks as assessed by 5-repetition Sit-to-stand (STS) test | It will be administered a total of 3 times during the whole study, including the beginning and end of the 12-week intervention, and the end of the 12-week follow up.
  A test that measures the time require to complete five consecutive sit-to-stand to-sit cycle as quickly as possible timed using a stop watch. Participants will be tested barefoot on a firm mat and the starting position with hip flexed at 90 degree and knee flexed at 105 degree. The ICCs of intra-session reliability and test-retest reliability were 0.95 and 0.99 respectively. The convergent validity was supported by significant correlation with isometric muscle strength, scores of Gross Motor Function Measure, and gait function (r or rho = 0.45-0.78).
Change from baseline in Body Function/Structure at 12 weeks and 24 weeks as assessed by Revised Dimensions of Mastery Questionnaire (DMQ 18) - Chinese version | It will be administered a total of 3 times during the whole study, including the beginning and end of the 12-week intervention, and the end of the 12-week follow up.
  The Revised Dimensions of Mastery Questionnaire (DMQ 18) - Chinese version: was used to measure both instrumental and expressive aspects of mastery motivation by caregiver report. There are 7 scales (cognitive/object persistence, gross motor persistence, social mastery motivation with adults, social mastery motivation with children/peers, mastery pleasure, negative reactions to challenge in mastery situations, and general competence) and Likert scale items rated 1-5 (from not at all like this child to exactly like this child). The higher score means the motivated performances are more like the child's behaviors. The DMQ 18 contained four parallel age-related versions for children aged 6 months to 19 years (infant, preschool, school-age rated by adults, and school-age self-report). The DMQ 18 show good internal consistency (.72-.96). The intra- and inter-rater reliability were acceptable for the DMQ18 (ICCs=0.61-0.87).
Change from baseline in General Development at 12 weeks and 24 weeks as assessed by The Bayley Scales of Development | It will be administered a total of 3 times during the whole study, including the beginning and end of the 12-week intervention, and the end of the 12-week follow up.
  An internationally recognized set of standardized developmental tests involves play and parental questionnaires. The Bayley has subsets of tests for motor (fine and gross), language (receptive and expressive), and cognitive development, ages from 0-3 years old.
Change from baseline in General Development at 12 weeks and 24 weeks as assessed by The Affordances in the Home Environment for Motor Development (AHEMD) | It will be administered a total of 3 times during the whole study, including the beginning and end of the 12-week intervention, and the end of the 12-week follow up.
  AHEMD is a reliable and valid assessment to assess the quality and quantity of motor development opportunities in the home during early childhood. Age-related AHEMD questionnaires were developed (3-to-18 months; and 18-to-42 months) and translated into four different languages: English, Chinese Portuguese, and Spanish. Test-retest reliabilities for AHEMD-Toddler-C were adequate (0.46~0.93). For convergent validity, the correlation coefficients between AHEMD and HOME were 0.44.
Change from baseline in Participation level at 12 weeks and 24 weeks as assessed by The Goal Attainment Scale (GAS) | It will be administered a total of 3 times during the whole study, including the beginning and end of the 12-week intervention, and the end of the 12-week follow up.
  GAS is a family-centered, criterion-referenced and responsive tool. There are 5 possible outcomes: a score of 0 means the child has attained the goal, whereas scores of -2 and -1 represent lower than expected performance and +1 and +2 are higher than expected performance. The Likert scale is used. The higher score means better achievements. It has excellent inter-rater agreements with inter-class correlations of 0.90 or above. GAS was shown to correlate strongly with other measures that showed change, and it discriminated between lower and higher functional or QOL status.
Physical Activity for Exploration as assessed by the number of counts recorded from the accelerators wearing on both wrists and the hip | The socialization behaviors will be followed for the duration of implementing the intervention phase, an expected average of 12 weeks.
  Each week the participant wears the accelerometers on both wrists and the hip during the 1 hour videotaping session, including 30-minute driving and 30-minute natural play. The accelerometers code the physical activity for driving and playing. Combining with the results from videotapes, this data enables us to understand the frequency and duration of bimanual use in different activities (i.e., manual exploration).
Change from baseline in Parents' Perception at 12 weeks and 24 weeks as assessed by Parenting Stress Index (PSI) | It will be administered a total of 3 times during the whole study, including the beginning and end of the 12-week intervention, and the end of the 12-week follow up.
  PSI is a tool that was designed to measure the overall level of parenting stress experienced by parents of children between the ages of one month and twelve years. PSI showed very good reliability (from parent : .55-.80). The validity was well established (factorial validity: 41% of variance on child section accounted for by 6 factors; 44% on Parent section by 7 parent factors).
Change from baseline in Parents' Perception at 12 weeks and 24 weeks as assessed by self-developed questionnaires | It will be administered a total of 3 times during the whole study, including the beginning and end of the 12-week intervention, and the end of the 12-week follow up.
  A set of self-developed questionnaires from the previous studies will be revised and used at T1, T2 and T3 to examine parental perceptions on the training programs and children's capabilities.

CONTACTS AND LOCATIONS:
Overall Officials: Hsiang-Han Huang, ScD, Principal Investigator — Chang Gung University
Locations (1):
- Chang Gung University, Taoyuan, Taoyuan County, Taiwan